CLINICAL TRIAL: NCT02937467
Title: Evaluation of Shear Wave Elastography in the Diagnosis and Management of Thyroid Nodules in Chinese Population: A Prospective, Multicenter Study
Brief Title: The Multi-Center Study of Shear Wave Elastography on Thyroid Nodules
Status: Available | Type: Expanded Access
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Yan, chief director, Peking University Cancer Hospital & Institute
Other Study IDs: SHSY-IEC-3.0/15-78/01
Record Dates: First submitted 2016-10-15; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Thyroid Nodules
Keywords: SWE; diagnosis
MeSH Terms: conditions — Thyroid Nodule; Disease

INTERVENTIONS:
Device: SWE — a novel ultrasound-based elastographic method, a new real-time, quantitative, operator-independent, and reproducible technique

SUMMARY:
The incidence rates of thyroid cancers have increased in the past decade. Additionally, up to 68% of people have thyroid nodules. Consequently, a precise evaluation of thyroid nodules is very important and can avoid unnecessary biopsy of benign nodules. Shear wave elastography(SWE), a novel ultrasound-based elastographic method, is a new real-time, quantitative, operator-independent, and reproducible technique. Briefly, shear wave elastography uses a radiation force produced by an ultrasonic beam to stress tissues and ultrafast sonographic tracking techniques to measure the speed of shear waves. Based on the Young modulus formula, tissue elasticity can be derived from the shear wave propagation speed, and a real-time color-coded elastogram can be displayed, showing softer tissue in blue and stiffer tissue in red.

There are lots of research confirmed that SWE has a certain value in the diagnosis of thyroid carcinoma. These studies include prospective studies and retrospective studies, but both belong to a single center study. It has not been applied to the study of the multicenter of thyroid disease.

The main purpose of the study is to assess the performance of SWE for identification of benign and malignant thyroid nodules and calculate the optimal cutoff value for each parameter in multicenter study; the secondary purpose is to evaluate the application value of SWE for uncertain nodules by FNA.

DETAILED DESCRIPTION:
SWE can prove the diagnostic performance in the differentiation of benign and malignant thyroid lesions

1. Main purpose

   1. to assess the performance of SWE for identification of benign and malignant thyroid nodules in multicenter study;
   2. calculate the optimal cutoff value for each parameter in multicenter study
2. Secondary purpose to evaluate the application value of SWE for uncertain nodules by FNA.

ELIGIBILITY:
Inclusion Criteria

1. the size of the lesion is between 0.5～4cm
2. the solid components in the lesion>50%；
3. all patients perform FNA or surgery in one month after SWE examination

Exclusion Criteria:

1. patients who are unwilling or unable to provide informed consent
2. Woman who is pregnant or breastfeeding;
3. Thyroid nodules with calcified which is beyond 1/2 diameter of lesion
4. patients who have history of surgery、FNA or thermal ablation in ipsilateral thyroid
5. patients who have serious cardiopulmonary diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: yan kun, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute; xu huixiong, Doctor, Principal Investigator — Shanghai 10th People's Hospital

REFERENCES:
- [Background] Berg WA, Cosgrove DO, Dore CJ, Schafer FK, Svensson WE, Hooley RJ, Ohlinger R, Mendelson EB, Balu-Maestro C, Locatelli M, Tourasse C, Cavanaugh BC, Juhan V, Stavros AT, Tardivon A, Gay J, Henry JP, Cohen-Bacrie C; BE1 Investigators. Shear-wave elastography improves the specificity of breast US: the BE1 multinational study of 939 masses. Radiology. 2012 Feb;262(2):435-49. doi: 10.1148/radiol.11110640. PMID 22282182
- [Background] Monpeyssen H, Tramalloni J, Poiree S, Helenon O, Correas JM. Elastography of the thyroid. Diagn Interv Imaging. 2013 May;94(5):535-44. doi: 10.1016/j.diii.2013.01.023. Epub 2013 Apr 25. PMID 23623210
- [Background] Xu JM, Xu XH, Xu HX, Zhang YF, Zhang J, Guo LH, Liu LN, Liu C, Zheng SG. Conventional US, US elasticity imaging, and acoustic radiation force impulse imaging for prediction of malignancy in thyroid nodules. Radiology. 2014 Aug;272(2):577-86. doi: 10.1148/radiol.14132438. Epub 2014 Apr 2. PMID 24689885
- [Background] Park AY, Son EJ, Han K, Youk JH, Kim JA, Park CS. Shear wave elastography of thyroid nodules for the prediction of malignancy in a large scale study. Eur J Radiol. 2015 Mar;84(3):407-412. doi: 10.1016/j.ejrad.2014.11.019. Epub 2014 Nov 27. PMID 25533720
- [Result] Shiina T, Nightingale KR, Palmeri ML, Hall TJ, Bamber JC, Barr RG, Castera L, Choi BI, Chou YH, Cosgrove D, Dietrich CF, Ding H, Amy D, Farrokh A, Ferraioli G, Filice C, Friedrich-Rust M, Nakashima K, Schafer F, Sporea I, Suzuki S, Wilson S, Kudo M. WFUMB guidelines and recommendations for clinical use of ultrasound elastography: Part 1: basic principles and terminology. Ultrasound Med Biol. 2015 May;41(5):1126-47. doi: 10.1016/j.ultrasmedbio.2015.03.009. Epub 2015 Mar 21. PMID 25805059